CLINICAL TRIAL: NCT04026308
Title: Written Safety Planning vs the Safety Net App: A Prospective Randomized Pilot Trial
Brief Title: Written vs Electronic Safety Planning Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 239731
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Suicidal Ideation; Suicide Attempt; Mental Health
Keywords: Suicide; Suicide Prevention; Safety Planning; Safety Net App
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Psychological Well-Being; Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Safety Plan (No Intervention): Participants will complete a traditional written suicide safety plan.
- Electronic Safety Plan (Experimental): Participants will complete a suicide safety plan in the Safety Net app using a tablet.
  Interventions: Other: Safety Net App

INTERVENTIONS:
Other: Safety Net App — The Safety Net app is an electronic version of a safety plan and it is available for download in Apple's App Store. A preview of the app is available at: https://apps.apple.com/us/app/stanley-brown-safety-plan/id695122998. This app is owned by Two Penguins Studios, LLC. It was developed in partnership with the New York State Office of Mental Health. Unlike the paper version, the Safety Net app allows participants to email a copy of their safety plan to whomever they wish. It also allows patients to dial 911 or the National Suicide Prevention Lifeline from the app.
  Other Names: Stanley-Brown Safety Plan App
  Arms: Electronic Safety Plan

SUMMARY:
Safety planning is a brief, ED-feasible intervention which has been demonstrated to save lives and has been universally recommended by every recent expert consensus panel on suicide prevention strategies. In one popular version of the safety plan developed by Stanley et al, the patient is encouraged to write out the following items: identifying personal signs of a crisis; helpful internal coping strategies; social contacts or settings which may distract from a crisis; using family members or friends for help when in crisis; mental health professionals who can be contacted when in crisis; and restricting access to lethal means.

This study aims to find out how valuable an electronic safety plan is compared to a traditional paper safety plan. People who are visiting the emergency department for thoughts of self-harm will be asked to participate.

DETAILED DESCRIPTION:
This project has 3 aims: (1) Will ED patients with suicidal ideation/attempt accept coaching on safety planning from non-clinical personnel (i.e., medical students or peer supporters); (2) Are these safety plans of high-enough quality for clinical personnel; and finally, (3) Will ED patients with suicidal ideation/attempt complete safety plans electronically?

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for suicidal ideation (SI) or after a suicide attempt to the UAMS ED
* Willingness to engage in safety planning with trained non-clinical staff
* Have not already filled out a safety plan at the current visit

Exclusion Criteria:

* <18 or >89 years of age
* Incarcerated or in police custody
* Non-English-speaking or Non-English-writing (as translators will not be available for this study)
* Critically-ill (or appear to be critically-ill)
* Intoxicated with alcohol or other substance(s)
* ED staff objection to patient enrollment in study
* Unwilling or unable to complete the safety plan electronically
* Unwilling or unable to use a tablet device to complete the safety plan
* Unwilling or unable to show/email the safety plan to clinical and research staff

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Wilson, M.D., Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Written Safety Plan | Electronic Safety Plan
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Written Safety Plan | Electronic Safety Plan | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 40 [21 to 69] | 39 [21 to 56] | 40 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: The number of patients approached who agree to allow trained non-clinical staff to assist with safety planning.
Time Frame: Up to 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Written Safety Plan | Electronic Safety Plan
Number analyzed (Participants) | 14 | 16
Participants | 14 | 16

2. Primary Outcome: Length of Stay
Description: The length of stay in the ED for patients approached who agree to allow trained non-clinical staff to assist with safety planning.
Time Frame: Up to 12 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Written Safety Plan | Electronic Safety Plan
Number analyzed (Participants) | 14 | 16
minutes | 250 [12 to 626] | 288 [13 to 978]

3. Primary Outcome: Satisfaction With Safety Planning
Description: Evaluate patient satisfaction with safety planning. This will be assessed by having the patient rate their experience with the safety planning process on a 7-point Likert scale (1 - strongly disagree; 2 - disagree; 3 - moderately disagree; 4 - neutral; 5 - moderately agree; 6 - agree; 7 - strongly agree). A Likert scale measures how much someone disagrees or agrees with a particular statement.
Time Frame: Up to 12 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Written Safety Plan | Electronic Safety Plan
Number analyzed (Participants) | 14 | 16
units on a scale | 5.29 [3 to 7] | 5.31 [4 to 7]

ADVERSE EVENTS:
Time Frame: Through participant's ED visit at enrollment, usually <1 day
Description: collected via REDCap
Arm/Group | Written Safety Plan | Electronic Safety Plan
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT04026308/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT04026308/ICF_001.pdf